CLINICAL TRIAL: NCT03111602
Title: Increase of Prostaglandin E2 in Reversal of Ductal Constriction After Dietary Restriction of Polyphenols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Izabele Vian, Principal Investigator / Dietitian, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18592013000005333
Record Dates: First submitted 2017-03-29; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy Complications
Keywords: polyphenols; pregnant; fetal ductal constriction; prostaglandin E2
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: Clinical trial with a healthy group as comparator.
Who Masked: Care Provider, Investigator
Masking Description: Researchers were blinded to the allocation data of pregnant women in the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): The interventional group was submitted to dietary orientation to restrict polyphenol-rich foods
  Interventions: Other: restrict polyphenol-rich foods
- control group (No Intervention): healthy group as comparator

INTERVENTIONS:
Other: restrict polyphenol-rich foods — dietary orientation to restrict polyphenol-rich foods
  Arms: interventional group

SUMMARY:
INCREASE OF PROSTAGLANDIN E2 IN REVERSAL OF DUCTAL CONSTRICTION AFTER DIETARY RESTRICTION OF POLYPHENOLS.

Clinical trial with a healthy group as comparator. The interventional group was made up of third-trimester mothers whose single fetuses had ductal constriction, excluding those exposed to NSAID, and the control group only by third-trimester normal fetuses. The interventional group was submitted to dietary orientation to restrict polyphenol-rich foods and both groups answered a food frequency questionnaire after fetal Doppler-echocardiographic examination and blood draw for PGE2 levels analysis. After two weeks, the women were again submitted to fetal echocardiogram, dietary assessment and blood draw.

DETAILED DESCRIPTION:
INCREASE OF PROSTAGLANDIN E2 IN REVERSAL OF DUCTAL CONSTRICTION AFTER DIETARY RESTRICTION OF POLYPHENOLS.

Fetal ductal constriction is a clinical situation with high morbidity and potential mortality. Patency the fetal ductus arteriosus (DA) depends on circulating prostaglandin (PG), which is produced by the cyclooxygenase (COX) pathway during inflammatory response(1) and from the third trimester of pregnancy on, is physiologically released. COX-inhibiting substances, such as nonsteroidal anti-inflammatory drugs (NSAIDs), can interfere with PG metabolism and induce constriction of the DA. To treat or prevent DA constriction, it is therefore important to reduce fetal exposure to drugs that may interfere with prostaglandin biosynthesis, such as natural anti-inflammatory drugs and polyphenol-rich foods.

Polyphenols, the most abundant antioxidants present in the diet, are widely distributed in vegetable foods. One of the possible mechanisms to explain their activity is inhibition of synthesis and release of inflammatory mediators. However, clinical studies investigating the effect of polyphenols on inflammatory responses are inconclusive and, in most cases, only evaluate clinical outcomes. The role of polyphenols on the inflammatory response, and associated modifications of the plasma concentration of PGE2 in pregnant women, has not yet been studied.

Despite the potential benefits of a diet rich in polyphenols, a high consumption of these substances in the third trimester of pregnancy may reduce plasma levels of PGE2 and result in DA constriction,so that a restriction in their ingestion during this period is already recommended.This functional problem has high prevalence and may result in severe fetal and neonatal complications. These considerations raised the hypothesis that reversal of fetal ductal constriction after maternal restriction of polyphenol-rich foods is accompanied by increased in prostaglandin E2 levels. Demonstration of this effect would represent an advancement in knowledge and might result in changes in dietary guidance during pregnancy and prevention of perinatal complications, with potential impact in terms of public health.

The aim of this study was to test the hypothesis that reversal of fetal ductal constriction in the third trimester of pregnancy, after maternal restriction of polyphenol-rich foods, is accompanied by increased plasma levels of prostaglandin E2.

ELIGIBILITY:
Inclusion Criteria

* Pregnancy with diagnosis of fetal ductal constriction
* Single fetus
* gestational age from 28 weeks

Exclusion Criteria

* cardiac malformations
* restricted intrauterine growth
* increased nuchal translucency
* present or suspected chromosomal disorders
* signs of any type of hydrops fetalis
* pregnancy
* hypertension
* diabetes mellitus
* structural or functional cardiac disorders
* current use of nonsteroidal anti-inflammatory drugs, steroids, antidepressants, illicit drugs, alcohol or smoking
* multiple pregnancy
* having received previous nutritional guidance in relation to restricted intake of polyphenol-rich foods

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant: third-trimester mothers
Enrollment: 75 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Plasma levels of prostaglandin E2 (PGE2) | baseline and two weeks
  PGE2 was quantified by capture ELISA. The measurements were obtained through 4-parameter linear regression (Excel, Microsoft), and data were expressed in picograms of protein per milliliter (pg/mL).

SECONDARY OUTCOMES:
Consumption of foods rich in Total Polyphenols (TP) | baseline and two weeks
  TP on the maternal diet were quantified using a Food Frequency Questionnaire (FFQ) validated for pregnant women. TP results after analysis of the dietary questionnaires were described in milligrams (mg)

OTHER OUTCOMES:
Diagnostic parameters of fetal ductus arteriosus constriction | baseline and two weeks
  The peak systolic, peak diastolic and end diastolic velocities (m/s) were determined. The pulsatility index of the ductus arteriosus was calculated automatically by the echocardiography system after manual tracing of the spectral curve, using the formula: (peak systolic velocity - diastolic peak velocity)/mean velocity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vian I, Zielinsky P, Zilio AM, Mello A, Lazzeri B, Oliveira A, Lampert KV, Piccoli A, Nicoloso LH, Bubols GB, Garcia SC. Development and validation of a food frequency questionnaire for consumption of polyphenol-rich foods in pregnant women. Matern Child Nutr. 2015 Oct;11(4):511-24. doi: 10.1111/mcn.12025. Epub 2013 Jan 15. PMID 23316751
- [Background] Momma K, Toyoshima K, Takeuchi D, Imamura S, Nakanishi T. In vivo constriction of the fetal and neonatal ductus arteriosus by a prostanoid EP4-receptor antagonist in rats. Pediatr Res. 2005 Nov;58(5):971-5. doi: 10.1203/01.pdr.0000182182.49476.24. PMID 16257930
- [Background] Zielinsky P, Piccoli AL Jr, Manica JL, Nicoloso LH, Vian I, Bender L, Pizzato P, Pizzato M, Swarowsky F, Barbisan C, Mello A, Garcia SC. Reversal of fetal ductal constriction after maternal restriction of polyphenol-rich foods: an open clinical trial. J Perinatol. 2012 Aug;32(8):574-9. doi: 10.1038/jp.2011.153. Epub 2011 Nov 3. PMID 22052330